CLINICAL TRIAL: NCT01617577
Title: Efficacy and Safety of Filgrastim as a Pro-Cognitive Agent in Alzheimer's Disease
Brief Title: Efficacy and Safety of Filgrastim in Alzheimer's Disease
Acronym: FFAD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADDF-GCSF
Record Dates: First submitted 2011-11-08; First posted 2012-06-12 (Estimated); Results first posted 2012-12-27 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-06

CONDITIONS: Alzheimer's Disease
Keywords: G-CSF; granulocyte colony stimulating factor; Filgrastim
MeSH Terms: conditions — Alzheimer Disease | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF (filgrastim) first phase (Experimental): Subjects assigned to this arm receive G-CSF for 5 days during the first phase of the study. At week 7 these subjects cross over to receive placebo injections for five days
  Interventions: Drug: G-CSF; filgrastim
- Placebo first phase (Placebo Comparator): Subjects assigned to this arm receive placebo injections daily for 5 days; after wk 7 they crossover to receive 5 daily injections of injections of G-CSF.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: G-CSF; filgrastim — The drug is administered s.c. at a dose of 10 microg/kg daily for 5 days
  Other Names: Neupogen; granulocyte colony stimulating factor (GCSF)
  Arms: G-CSF (filgrastim) first phase
Drug: Placebo — vehicle (D5W or 5% dextrose solution) is administered subcutaneously daily for 5 days
  Other Names: Vehicle (5% dextrose water or D5W)
  Arms: Placebo first phase

SUMMARY:
Filgrastim (G-CSF) is widely used for treatment of patients who have a deficiency of white blood cells. It is also routinely used to stimulate and mobilize stem/progenitor cells for bone marrow transplantation. In studies of thousands of healthy donor subjects treated with G-CSF, the side-effects profile has been reported to be mild and reversible. Currently, G-CSF is under investigation in clinical trials in Germany and the US that aim to enhance recovery from strokes and heart attacks. In animal studies, G-CSF has been observed to improve cognitive performance and to markedly reduce amyloid deposition in hippocampus and entorhinal cortex in a mouse model of Alzheimer's Disease (AD). Since this drug is being used safely in many people throughout the world, the investigators hypothesize that it will also be safe to give to patients with Alzheimer's disease and that it may improve some aspects of memory and thinking. The present pilot study has two goals or objectives: 1) to investigate the effects of a five day schedule of Filgrastim administration on cognitive function and 2) to assess its tolerability and safety in a small group (12 patients) with mild to moderate stage AD. Patients who are eligible for the study will be randomly assigned to one of two groups (n=6 per group). One group will receive a five-day course of Filgrastim injections and the other group of subjects will receive vehicle injections (solution without drug). At the end of the first phase of the study (week 8), the groups will cross over to receive either vehicle or Filgrastim as appropriate. In this way all subjects will have received the active medication by the end of the study. After the study is finished the investigators should know whether or not Filgrastim improves some aspects of thinking and memory. And the investigators should know whether or not it is safe to give this medication to patients with Alzheimer's disease. To ensure that the drug is safe, a Safety Monitoring Committee will oversee the entire study. They will review all laboratory data, including complete blood counts, serum chemistry, EKGs and adverse events.

DETAILED DESCRIPTION:
The study was originally designed to have two arms (GCSF first followed by placebo= Arm 1; placebo followed by GCSF=Arm2). Total length of study for each subject was 14 weeks, with crossover on week 7.

Linear regression models could not be used because of the small number of subjects; n = 5 in the first Arm who received G-CSF before crossover to the placebo phase and n = 3 in Arm 2 (who received placebo first before crossover to the G-CSF treatment phase). The general rule for the sample size required for regression analysis is n = 15 per covariate. Therefore, comparison of the final cognitive scores on visit 5 (week 14) were compared to scores at baseline (visit 1) for all subjects (n = 8) using the Wilcoxon signed rank test. Plasma cytokine changes were plotted to compare effects following G-CSF to that following placebo, regardless of the order of treatment. Wilcoxon sum rank test was used to test differences between G-CSF treatment and placebo treatment at specific intervals after treatment. Statistical Package for the Social Sciences (SPSS Version 19) was used for all data analysis.

ELIGIBILITY:
Inclusion Criteria:

* People with probable AD (by NINDS/ADRDA criteria) who are likely to be testable at the conclusion of the study period, and who do not have concurrent medical conditions or medications that might influence cognitive testing or that would increase the risk of treatment
* The participants will have a Min Mental State Examination score of between 10 and 24
* stable medical condition and stable medications for 3 months prior to screening
* study partner (spouse or caregiver) to accompany patient to all scheduled visits; able to complete baseline assessments
* physically acceptable for this study as confirmed by medical history, physical exam, neurological exam and clinical tests

Exclusion Criteria:

* clinically significant cardiac arrhythmia
* history of clinically significant stroke
* use of another investigational drug within 2 months of screening
* current evidence or history in the past 2 years of epilepsy, focal brain lesion, head injury with loss of consciousness or DSM-IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder alcohol or substance abuse; residence in a skilled nursing facility (but patients in assisted living facility are acceptable)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- USF/Byrd Alzheimer's Center, Tampa, Florida, United States

REFERENCES:
- [Background] Sanchez-Ramos J, Song S, Sava V, Catlow B, Lin X, Mori T, Cao C, Arendash GW. Granulocyte colony stimulating factor decreases brain amyloid burden and reverses cognitive impairment in Alzheimer's mice. Neuroscience. 2009 Sep 29;163(1):55-72. doi: 10.1016/j.neuroscience.2009.05.071. Epub 2009 Jun 14. PMID 19500657
- See also: Related Info — http://www.alzdiscovery.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- G-CSF First Phase: Subjects assigned to this arm receive G-CSF for 5 days during the first phase of the study. At week 7 these subjects cross over to receive placebo injections for five days
Period: Overall Study
Arm/Group | G-CSF First Phase | Placebo First Phase
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | G-CSF First Phase | Placebo First Phase | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 2 | 2 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 71.6 (3.8) | 75.2 (3.1) | 72.3 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Measures Incluing ADAScog, Selected CANTABS Tests (Paired Associate Learning (PAL)and PAL )
Description: Scores from each of the cognitive assessments:
  mean ADAScog: a decrease in total score units = improvement, min=0 max=31 mean PAL (memory): an increase in score = improvement, min= 0 max=12 mean PAL (total trial adj): a decrease in score = improvement,
Time Frame: Baseline and 2wk and 4 wk after Rx;
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- G-CSF: All participants received G-CSF either in the first or second phase of the crossover
- Placebo: All participants received placebo either in the first or second phase of crossover
Arm/Group | G-CSF | Placebo
Number analyzed (Participants) | 8 | 8
units on a scale
  ADAScog Baseline | 22.25 (2.49) | 22.25 (2.49)
  ADAScog 2wk post Rx | 20.5 (1.67) | 17.75 (2.67)
  ADAScog 4wks post Rx | 21.5 (2.507) | 20.125 (2.14)
  PALmem baseline | 2.75 (0.59) | 2.75 (0.59)
  PALmem 2wk post Rx | 4.14 (0.857) | 3.75 (1.06)
  PALmem 4wk post RX | 5.50 (1.477) | 4.75 (0.881)
  PAL (tot trial adj) baseline | 33.87 (3.02) | 33.87 (3.02)
  PAL (tot trial adj) 2wk post Rx | 28.48 (6.16) | 33.62 (4.26)
  PAL(tot trial adj) 4wk post RX | 24.45 (5.36) | 30.62 (3.02)

2. Primary Outcome: Cognitive Measures Incluing ADAScog, Selected CANTABS Tests (Paired Associate Learning (PAL)and PAL )
Description: Scores from each of the cognitive assessments:
  mean ADAScog: a decrease in total score units = improvement, min=0 max= mean PAL (memory): an increase in score = improvement, mean PAL (total trial adj): a decrease in score = improvement,
Time Frame: Baseline and final visit (14 wks)
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- G-CSF and Placebo: All participants received G-CSF and placebo in crossover order
Arm/Group | G-CSF and Placebo
Number analyzed (Participants) | 8
units on a scale
  ADAScog Baseline | 24 (2.86)
  ADAScog 14wks post Rx | 20.37 (2.25)
  PALmem baseline | 2.85 (0.67)
  PALmem 14wk post RX | 5.17 (1.41)
  PAL (tot trials adj) baseline | 33.88 (3.003)
  PAL (tot trials adj) 14wk post RX | 30. (3.65)
Statistical Analysis 1: Comparison: G-CSF and Placebo; ADAScog scores at baseline vs final visit (wk 14); null hypothesis is there is no difference between scores; Test type: Superiority or Other; p = 0.36, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test
Statistical Analysis 2: Comparison: G-CSF and Placebo; PAL(mem) at baseline and 14 wk (final visit): null hypothesis is thereis no difference in score; Test type: Superiority or Other; p = 0.058, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test
Statistical Analysis 3: Comparison: G-CSF and Placebo; PALtot trials adj at baseline vs 14wk (final visit); Test type: Superiority or Other; p = 0.034, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test

ADVERSE EVENTS:
Groups:
- Placebo: subjects who received placebo in either phase of the study
- G-CSF: participants who received GCSF injecitons during first or second phase
Arm/Group | Placebo | G-CSF
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | G-CSF (N=8)
headache (Nervous system disorders) | 1 (1) | 1 (1) — all headaches occured after lumbar puncture regardless of GCSF or placebo treatment
generalized aches (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) — relieved in all subjects with non-steroidal anti-inflammatory agents (tyelone or motrin)
back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
nausea (Nervous system disorders) | 1 (1) | 1 (1)
visual hallucinations (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No